CLINICAL TRIAL: NCT00176137
Title: Cisplatin/Etoposide Followed by Twice-Daily Chemoradiation (hfRT/CT) Versus Cisplatin/Etoposide Alone Before Surgery in Stage III Non-Small Cell Lung Cancer. A Phase III Trial of the German Lung Cancer Cooperative Group (GLCCG)
Brief Title: Preoperative Twice Daily Chemoradiation in Addition to Chemotherapy Prior to Surgery in Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: University Hospital Muenster (Other); Lung Clinic Hemer (Other); Kreiskrankenhaus Diekholzen (Unknown); University Hospital, Saarland (Other); FLT Berlin / Buch (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLCCG01/95; German Cancer Aid
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: multimodality treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Procedure: preoperative radiochemotherapy

SUMMARY:
Patients are randomized to (arm A) 3 cycles of cisplatin/etoposide, followed by hyperfractionated radiotherapy (hfRT)with concurrent carboplatin and vindesine then surgery and, if no or R1/2-resection, additional hfRT versus (arm B) 3 cycles of cisplatin/etoposide, followed by surgery and then RT.

The primary endpoint was progression free survival (PFS). With 500 patients evaluable an improvement of median PFS from 10 to 14 months could be detected.

DETAILED DESCRIPTION:
Patients are randomized to (arm A) 3 cycles of cisplatin 55 mg/m2 (d 1 + 4)/etoposide 100 mg/m2 (d 1-4), followed by hyperfractionated radiotherapy (hfRT; 45 Gy, 2x1.5 Gy/d) with concurrent carboplatin (100 mg/m2) and vindesine (3 mg) (d 1, 8, 15), then surgery and, if no or R1/2-resection, additional hfRT (24 Gy; 2x1.5 Gy/d) versus (arm B) 3 cycles of cisplatin 55 mg/m2 (d 1 + 4)/etoposide 100 mg/m2 (d 1-4),followed by surgery and then RT (1.8 Gy/d) with 54 Gy or, if no or R1/2-resection, 68.4 Gy.

The primary endpoint was progression free survival (PFS). With 500 patients evaluable an improvement of median PFS from 10 to 14 months could be detected.

(University of Münster was the lead sponsor; as the trial was implemented in clinicaltrials.gov by the principal investigator after he had moved to University of Heidelberg this account is announced above)

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer proven by histology
* stage IIIA / stage IIIB
* mediastinoscopy
* performance score ECOG 0,1
* predicted postoperative FEV 1 > 1.0 l

Exclusion Criteria:

* small cell lung cancer
* cardiac disability (NYHA III/IV)
* prior radio- or chemotherapy
* pregnancy
* other malignancy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1995-10; Study Completion 2005-09

PRIMARY OUTCOMES:
Progression free survival

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thomas, Prof. / MD, Study Chair — Current affiliation: Thoraxklinik am Universitätsklinikum Heidelberg

REFERENCES:
- [Derived] Kreuter M, Kropff M, Fischaleck A, Junker K, Gerss J, Heinecke A, Lindermann M, Reinmuth N, Berdel WE, Mesters RM, Thomas M. Prognostic relevance of angiogenesis in stage III NSCLC receiving multimodality treatment. Eur Respir J. 2009 Jun;33(6):1383-8. doi: 10.1183/09031936.00121108. Epub 2009 Feb 12. PMID 19213790
- [Derived] Thomas M, Rube C, Hoffknecht P, Macha HN, Freitag L, Linder A, Willich N, Hamm M, Sybrecht GW, Ukena D, Deppermann KM, Droge C, Riesenbeck D, Heinecke A, Sauerland C, Junker K, Berdel WE, Semik M; German Lung Cancer Cooperative Group. Effect of preoperative chemoradiation in addition to preoperative chemotherapy: a randomised trial in stage III non-small-cell lung cancer. Lancet Oncol. 2008 Jul;9(7):636-48. doi: 10.1016/S1470-2045(08)70156-6. Epub 2008 Jun 24. PMID 18583190